CLINICAL TRIAL: NCT07191925
Title: An Evaluation of "Growing Healthy Places: Mississauga"
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Collaborators: Novo Nordisk A/S (Industry); Delivery Associates (Unknown); Ophea (Unknown); 8 80 Cities (Unknown); The Behavioural Insights Team (Other)
Responsible Party: Principal Investigator, Karen Patte, PhD, Associate Professor, Health Sciences, Brock University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB24-273
Record Dates: First submitted 2025-09-08; First posted 2025-09-25 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Quality of Life (QOL); Physical Activity; Diet Quality; Obesity &Amp; Overweight; Body Esteem; Community
Keywords: health behavior; child health; multi-level; community intervention
MeSH Terms: conditions — Motor Activity; Obesity; Overweight; Health Behavior

STUDY DESIGN:
Intervention Model Description: Clustered intervention: participants within 22 school clusters (10 intervention, 12 control) from 11 unique neighborhoods assigned to either intervention or control for the study duration
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receive a community co-designed package of multi-level, multi-component interventions targeting physical activity and diet
  Interventions: Behavioral: Community Co-designed Physical Activity and Diet Intervention Package
- Control Group (No Intervention): Usual school and community practices with no interventions from the study

INTERVENTIONS:
Behavioral: Community Co-designed Physical Activity and Diet Intervention Package — A package of 4-6 diet and physical activity interventions selected from a long-list of potential interventions and adapted to the unique school and neighborhood context via consultation with community stakeholders. Intervention packages are multi-level (i.e. targeting at least two of individual, external and structural environments), target elements of both diet and physical activity, and are health equity oriented in terms of both access and improvement. Long-list potential interventions include items related to school intramural programming, active transport, health education, community recreational programming, and structural/public space design improvements.
  Arms: Intervention Group

SUMMARY:
The goal of this intervention study is to learn if community co-designed activities to improve diet and physical activity can impact the health of children ages 6-13 in Mississauga, Canada. The main questions it aims to answer are:

1. Do the community co-designed interventions improve health-related quality of life of children after one year and two years?
2. Do the community co-designed interventions improve the physical activity and eating behaviors of children after one year and two years?

Ten intervention and 12 control schools will take part in this study. The schools were recruited from the Mississauga area using an application process. Selection and group assignment involved a multi-stage process with initial randomization followed by manual adjustment (to balance groups on key observable characteristics and respond to stakeholder concerns about spillovers and implementation feasibility).

Researchers will compare students in schools that receive the interventions to students in schools that receive no interventions to see if the interventions improve health-related quality of life, increase physical activity and improve eating behaviors.

Participants will:

* attend participating elementary or middle schools (in either intervention neighborhoods or control neighborhoods)
* complete an anonymous questionnaire about their wellbeing, physical activity, and eating behaviors at baseline, after one year, and after two years
* potentially participate in school and community programs (if in an intervention school neighborhood)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained by the child's parent or legal guardian before any study-related activities
* Aged 6-13 years (both 6 and 13 allowed) at the time of signing consent
* Enrolled in Grades 3-8 in one of the participating schools at the time of data collection

Exclusion Criteria:

* Parent(s) or legal guardians do not provide fully informed consent
* Parent(s) or legal guardians withdraw their consent for their child participating in the research
* Child does not agree to participate on the data collection day

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4900 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Health-related Quality of Life as assessed by KIDSCREEN-10 index | Baseline, one-year follow-up, two-year follow-up.
  Health-related quality of life will be proxied by the KIDSCREEN-10 scale, which is developed from 27-item KIDSCREEN-27 scale and assesses health-related quality of life on five dimensions: physical, psychological, autonomy and parent relations, peers and social support, school environment. Each item uses a 5-point Likert-style response based on how strong the respondent is feeling or the frequency of doing / feeling things over the last week.
  KIDSCREEN instruments were originally designed for ages 8-18 but have been validated in ages 6-18. Item wording is slightly adapted for typical Canadian phrasing.
  Responses to each item are coded 1-5, items scores are summed, and the total score is linearly transformed to a 0-100 scale. A higher score corresponds to a higher health-related quality of life.

SECONDARY OUTCOMES:
Average daily moderate-to-vigorous physical activity (MVPA) | Baseline, one-year follow-up, two-year follow-up
  Daily minutes of moderate-to-vigorous physical activity is measured using a single questionnaire item adapted from the Youth Health - Physical Activity & Sedentary Behavior Module questionnaire. The question that asks students to indicate the total time range in minutes spent doing moderate or vigorous physical activities the previous day (with examples provided). Provided time intervals are adjusted depending on the age of the participant to facilitate accurate recall. Total MVPA time is calculated by assuming the midpoint of the time interval.

OTHER OUTCOMES:
Total daily physical activity time including walking | Baseline, one-year follow-up, two-year follow-up
  Daily minutes of total physical activity will be measured using two items adapted from the Youth Health - Physical Activity & Sedentary Behavior Module questionnaire. Separate items ask students to indicate the total time range in minutes spent doing moderate-to-vigorous physical activities and spent walking during the previous day. Provided time intervals are adjusted depending on the age of the participant to facilitate accurate recall. Total physical activity time is calculated by summing the time from each item, assuming the midpoint of the time interval.
Average daily sedentary time (out-of-school recreational screen time) | Baseline, one-year follow-up, two-year follow-up
  Daily sedentary time, defined as out-of-school recreational screen time, will be measured using a single item adapted from the Youth Health - Physical Activity & Sedentary Behavior Module questionnaire. The question asks students to indicate the total time range in minutes spent sitting or lying down looking at a smartphone, tablet, computer, or TV outside of school during the previous day. Provided time intervals are adjusted depending on the age of the participant to facilitate accurate recall. Total sedentary time is calculated by assuming the midpoint of the time interval.
Estimated energy expenditure | Baseline, one-year follow-up, two-year follow-up
  Energy expenditure through physical activity is estimated as total kilocalories (kcal) burned during moderate-to-vigorous (MVPA) and non-MVPA physical activity time, based on total physical activity time indicated from survey responses. Energy expenditure in kcal/minute is the product of the MET (metabolic equivalent) x BMR (base metabolic rate), where MET is assumed to be 5.5 for MVPA activities and 3.0 for non-MVPA activities, and BMR is based on age- and sex-adjusted Schofield equations. Total daily energy expenditure is then estimated using a MET of 1.2 for non-physical activity time, which is estimated as 24 hours less physical activity time.
Global dietary recommendations score | Baseline, one-year follow-up, two-year follow-up
  Global dietary recommendations (GDR) score will be measured with an edited version of the Diet Quality Questionnaire (DQQ), which asks children whether they ate foods from each of 29 food groups in any of four meals (breakfast, lunch, dinner, snack) in the previous day. A simplified 16-food group version is used for children in grades 3-4. The total GDR is calculated based on sub-scores for consumption counts of food categories (fruits and vegetables, sugar-sweetened beverages, added sugars, saturated fats, fibre, starchy staples, dairy food, animal-source food).
Estimated energy intake | Baseline, one-year follow-up, two-year follow-up
  Energy intake is estimated as total kilocalories (kcal) consumed based on responses to each item in the Diet Quality Questionnaire. Each item is assigned an estimated unweighted average kcal intake for children across al food items mentioned within that item. Kcal values will be summed across all items and mealtimes indicated to produce a total estimated energy intake for the previous date.
Estimated net calories | Baseline, one-year follow-up, two-year follow-up
  Net calories is estimated in kcal/day for each participant as total estimated energy expended minus total estimated energy intake
Experiences of food insecurity (Gr5-8 only) | Baseline, one-year follow-up, two-year follow-up
  Experience of food insecurity within the home context will be measured using a single question item asking how often in the last month the participant worried about running out of food to eat at home, with pre-specified frequency response options ranging from never to every day. These questions are only asked to participants in grades 5 to 8.
Participation in school food program (Gr5-8 only) | Baseline, one-year follow-up, two-year follow-up
  Participation within a school food program will be measured using a single question item asking how often in the last month the participant ate food that was provided by the school for free (such as a breakfast, lunch, or snack), with pre-specified frequency response options ranging from never to every day. These questions are only asked to participants in grades 5 to 8.
Physical literacy (Gr5-8 only) | Baseline, one-year follow-up, two-year follow-up
  Physical literacy (defined as the competence, confidence, and motivation to participate in a variety of sports and physical activities) will be measured using two questionnaire items adapted from the PLAY self tool. The items ask participants to indicated their level of agreement on a 4-point Likert-style scale to two statements regarding feeling confident when doing physical activities, and feeling happier when being active. These questions are only asked to participants in grades 5 to 8.
Perception of school physical activity context (Gr5-8 only) | Baseline, one-year follow-up, two-year follow-up
  Perceptions/experiences of physical activity within the school context will be examined through a single questionnaire item related to feeling welcome when doing physical activity at school. The item ask participants to indicated their level of agreement on a 4-point Likert-style scale. This question is only asked to participants in grades 5 to 8.
Sense of belonging in school | Baseline, one-year follow-up, two-year follow-up
  Sense of belonging within one's school will be assessed using items capturing various aspects of school connection. Each item uses a 5-point Likert-style response based on how strong the respondent is feeling or the frequency of doing / feeling things over the last week. Two items adapted from the KIDSCREEN-27 questionnaire will be asked of all participants: feeling happy at school and having fun. Two additional optional items related to feeling safe at school and feeling a part of one's school will be asked among participants in grades 5-8 only. A total sense of belonging score will be calculated by summing available item responses based on participant grade.
Body image and body appreciation (Gr5-8 only) | Baseline, one-year follow-up, two-year follow-up
  Positive body image and body appreciation will be measured using items from the Body Appreciation Scale-2 for Children, which generates a sum score based on 8 items related to positive feelings and attitudes toward one's body. These optional measures will only be asked among participants in grades 5-8.
Sense of belonging in one's community (Gr5-8 only) | Baseline, one-year follow-up, two-year follow-up
  Sense of belonging within one's community will be assessed using five items adapted from a community cohesion scale used in the Health Behavior of School-aged Children study. Items assess aspects of community trust, safety, support, communication, and facilities. Items are scored using a 5-point Likert scale for level of agreement and then summed to calculate a total community belonging score. These optional items will only be asked among participants in grades 5-8.
Intervention Reach: total people reached | Continuously throughout intervention phase: post-baseline to pre-two-year follow-up
  Total number of people reached by each intervention will collected by local delivery partners for each intervention and aggregated quarterly during the intervention delivery phase to determine the total across all interventions.
Intervention Reach: total children (0-18 years) reached | Continuously throughout intervention phase: post-baseline to pre-two-year follow-up
  Total number of children (0-18 years) reached by each intervention will collected by local delivery partners for each intervention and aggregated quarterly during the intervention delivery phase to determine the total across all interventions.
Intervention Reach: total target population reached (6-13 years) | Continuously throughout intervention phase: post-baseline to pre-two-year follow-up
  Total number target population (6-13 years) reached by each intervention will collected by local delivery partners for each intervention and aggregated quarterly during the intervention delivery phase to determine the total across all interventions.
Impact: Estimated change in BMI-z score | One-year follow-up, two-year follow-up
  Estimated impact on BMI is modelled using the PRIMEtime simulation model. Net calorie change (based on estimated net calories from questionnaire items) is translated into predicted changes in average body weight, which are then expressed as BMI z-scores.
Impact: Estimated change in incidence of cardiovascular disease | One-year follow-up, two-year follow-up
  Estimated impact on cardiovascular disease (CVD) incidence is modelled using the PRIMEtime simulation model. Predicted BMI changes are linked to risk equations for cardiovascular disease incidence and mortality, altering the projected disease burden.
Impact: Estimated change in incidence of Type 2 diabetes | One-year follow-up, two-year follow-up
  Estimated impact on Type 2 diabetes incidence is modelled using the PRIMEtime simulation model. Predicted BMI changes are input into established risk models for type 2 diabetes, altering projected onset and prevalence.
Impact: Estimated change in quality-adjusted life years (QALYs) | One-year follow-up, two-year follow-up
  Estimated impact on quality-adjusted life years (QALYs) is modelled using the PRIMEtime simulation model. Reductions in projected disease incidence and mortality are converted into gains in health-adjusted survival.
Impact: Estimated change in disability-adjusted life years (DALYs) | One-year follow-up, two-year follow-up
  Estimated impact on disability-adjusted life years (DALYs) is modelled using the PRIMEtime simulation model. The model estimates years of healthy life gained by reducing both premature death and years lived with disability.
Impact: Cost-effectiveness of interventions | One-year follow-up, two-year follow-up
  Cost-effectiveness of interventions is modelled using the PRIMEtime simulation model. Health care costs associated with each disease are combined with QALY/DALY projections to calculate incremental cost-effectiveness ratios (ICERs) and overall net monetary benefit.

CONTACTS AND LOCATIONS:
Locations (1):
- School Board, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be shared with global research collaborators (The Behavioural Insights Team, Oxford University). Novo Nordisk A/S will receive grouped data.
Supporting Information: Study Protocol